CLINICAL TRIAL: NCT07267689
Title: Performance and Safety Evaluation of a Hypertonic Seawater Aerosol Therapy Solution in Adults and Children With Upper Respiratory Tract Infection: a Prospective and Multicenter Study
Brief Title: Evaluation of a Hypertonic Seawater Aerosol Therapy Solution in Adults and Children
Acronym: AIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Gilbert (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAR-2022-0832
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Upper Resp Tract Infection; Rhinitis Acute; Rhinopharyngitis; Cold Symptom; Rhinitis Viral
Keywords: hypertonic seawater; upper respiratory tract infection (URTIs); inhalation; nebulization
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold; Nasopharyngitis; Respiratory Aspiration | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Pivotal clinical investigation Interventional, prospective, non-comparative, open, multicentric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient treated with 22‰ Hypertonic seawater solution, used as aerosol therapy for inhalati (Experimental): 5mL of 22‰ Hypertonic seawater per treatments, 14 treatments on 7 consecutive days
  Interventions: Device: Treatment (22‰ Hypertonic seawater aerosol therapy solution)

INTERVENTIONS:
Device: Treatment (22‰ Hypertonic seawater aerosol therapy solution) — Treatment twice a day for 7 consecutive days with 22‰ Hypertonic seawater aerosol therapy solution used in association with a nebulizer

SUMMARY:
The purpose of this study is to evaluate the tolerance, the performance and safety of this device, 22‰ Hypertonic seawater aerosol therapy solution in unidose container, to treat adult and peadiatric patients with of upper respiratory tract infection such as rhinopharyngitis, rhinitis, acute rhinosinusitis or cold.

The main questions it aims to answer are to assess if the 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation:

* improve nasal symptoms relief;
* improve sleep quality;
* improve mucus fluidizing;
* is safe and well tolerated.

The study is none comparative and will assess prospectively the symptomatic and functional benefits, the tolerance and the general safety of the medical device when used as an aerosol therapy solution, measured by change from baseline.

Treatments will be done at home and participants will be required to perform two on sites visits and to complete questionnaires and scales for 7 consecutive days from the treatment starting.

DETAILED DESCRIPTION:
Hypertonic seawater-based solution is a simple and well-known product. The performance of these solutions has been established in paediatric (infants, children), and in adult populations. The mode of action is based on the physical (mechanical) osmotic effect of the solution. Hypertonic saline induces an osmotic flow of water into the mucus layer, rehydrating the airway surface liquid and improving mucus clearance. Hypertonic saline also reduces viscosity and elasticity of mucus.

Hypertonic saline solution (seawater based or not) can be used for intranasal wash, or in association with a nebulization system as an aerosol therapy solution for inhalation. Inhalation via nebulization allows the formation of fine particles or liquid droplets in a gas.

In this study, 22‰ Hypertonic seawater solution, in unidose container, manufactured by Laboratoires Gilbert will be used as an aerosol therapy solution for inhalation in the treatment of URTIs such as rhinopharyngitis, rhinitis, acute rhinosinusitis or cold. The investigational medical device 22‰ Hypertonic seawater solution from Laboratoires Gilbert will be used in association with a nebulization system.

The purpose of this study is to evaluate the tolerance, the performance and safety of this device, 22‰ Hypertonic seawater aerosol therapy solution in unidose container, to treat adult and peadiatric patients with of upper respiratory tract infection such as rhinopharyngitis, rhinitis, acute rhinosinusitis or cold.

The main questions it aims to answer are to assess if the 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation:

* improve nasal symptoms relief;
* improve sleep quality;
* improve mucus fluidizing;
* is safe and well tolerated.

The study is none comparative and will assess prospectively the symptomatic and functional benefits, the tolerance and the general safety of the medical device when used as an aerosol therapy solution, measured by change from baseline.

Treatments will be done at home and participants will be required to perform two on sites visits and to complete questionnaires and scales for 7 consecutive days from the treatment starting.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subject voluntarily given informed consent to investigation participation in writing encompassing consent to data recording and verification procedures.
2. Minor subjects (7-17 years old) given informed assent to investigation participation in writing encompassing consent to data recording and verification procedures
3. Male and female subjects, aged from 2 years old;
4. Subject with URTIs such as rhinopharyngitis, rhinitis, acute rhinosinusitis or cold.
5. Subject willing to adhere to the requirements of the protocol, including availability for follow-up visits
6. Subject who is able to comply with the study requirements, at the Investigator's appreciation.
7. For minor (<18) subjects, parents/guardians willing and able to sign written consent

Exclusion Criteria:

1. Person with hypersensitivity to seawater
2. Subject who previously undergone bronchospasm
3. Children under 2 years of age
4. Pregnant and breastfeeding women
5. Onset of URTI symptoms > 48 hours
6. Subject known to have allergy to the components of the masks that is used with the inhalation device;
7. Subject with asthma;
8. Subject presenting infection or pathology of the inferior respiratory tracts;
9. Subject with chronic nasal obstruction (polypes)
10. Subject agrees to not used other saline solutions (irrigation), nasal spray, antihistamines, steroids, antipyretics, analgesic, antibiotics, decongestants, local antispectic, essential oil for nasal use and gel or nasal cream during study participation
11. Subject with drug or alcohol abuse
12. Subjects who is deprived for their freedom by administrative or legal decision
13. Subject living in a social or sanitary establishment.
14. Subject being in an exclusion period for a previous study or with a current or recent (<3 months) participation in another investigational study involving a drug or combined device with drug.
15. Other condition preventing the subject to participate the study in the investigator's opinion: subject deemed unreliable or incapable of understanding and complying with the study assessment or unrealistic expectations of treatment results.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
- Evaluate the performance of 22‰ Hypertonic seawater solution, used as aerosol therapy solution for inhalation, on the evolution of nasal symptom relief using the WURSS-21 questionnaire in minor patients from 14 years old and adults. | From Day 1 to Day 3
  Change in global WURSS-21 score as measured in the morning before treatment on Day 1 and Day 3 .
Evaluate the performance of 22‰ Hypertonic seawater solution, used as aerosol therapy solution for inhalation, on the evolution of nasal symptom relief using the WURSS-K questionnaire in minor patients from 4 to 13 years old. | From Day 1 to Day 3
  Change in global WURSS-K score as measured in the morning before treatment on Day 1 and Day 3.

SECONDARY OUTCOMES:
Evaluate the performance of 22‰ Hypertonic seawater solution, used as aerosol therapy solution for inhalation, on the evolution of nasal symptom relief using the WURSS-21 questionnaire in minor patients from 14 years old and adults. | Day 1, Day 2, Day 4, Day 5, Day 6, Day 7 and Day 8
  Change in global WURSS-21 score as measured in the morning before treatment at Day2, at Day 4, at Day 5, at Day 6, at Day 7 and at Day 8 compared to Day 1 (before treatment) as baseline.
Evaluate the performance of 22‰ Hypertonic seawater solution, used as aerosol therapy solution for inhalation, on the evolution of nasal symptom relief using the WURSS-K questionnaire in minor patients from 4 to 13 years old. | Day 1, Day 2, Day 4, Day 5, Day 6, Day 7 and Day 8
  Change in global WURSS-K score as measured in the morning before treatment at Day 2, at Day 4, at Day 5, at Day 6, at Day 7 and at Day 8 compared to Day 1 (before treatment) as baseline.
Assess the immediate benefit of 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation on nasal symptom relief. | Day 1, Day 3, Day 5 and Day 7
  Change in VAS (Visual Analog Scale) score before and immediately after treatment (nasal symptom relief).
Assess the proportion of patients that note an immediate benefit of 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation on nasal symptom relief. | Day 1, Day 3, Day 5 and Day 7
  Proportion of patients reporting improvement in nasal symptom relief (defined as a VAS increase of more than 3 points on a 10-point scale) immediately after treatment.
Assess the sustained benefit of 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation on nasal symptom relief. | Day 1, Day 3, Day 5 and Day 7
  Change in VAS (Visual Analog Scale) score before treatment and 3 hours post-treatment (nasal symptom relief).
Assess the proportion of patients that note a sustained benefit of 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation on nasal symptom relief during the day. | Day 1, Day 3, Day 5 and Day 7
  Proportion of patients reporting improvement in nasal symptom relief (defined as a VAS increase of more than 3 points on a 10-point scale) 3 hours post- treatment
Assess the benefit of 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation in improving sleep quality. | Day 1 before treatment, Day 2, Day 3, Day 5 and Day 7
  Improvement in sleep quality defined as a VAS score increase of more than 3 points on a 10-point scale, in the morning following evening treatment compared to baseline (assessment at Day 1 before treatment regarding the sleep quality during the night between Day 0 and Day 1).
Assess the proportion of patients reporting an improvement of sleep quality following evening treatment with the of 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation. | Day 1 before treatment, Day 2, Day 3, Day 5 and Day 7
  Proportion of patients reporting improvement in sleep quality (defined as a VAS increase of more than 3 points on a 10-point scale), in the morning following evening treatment with the device compared to baseline (assessment at Day 1 before treatment regarding the sleep quality during the night between Day 0 and Day 1)
Evaluate the performance of 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation on the improvement of mucus fluidizing | Day 1, Day 3, Day 5, Day 7
  Assess performance to improve mucus fluidizing (6-point Likert scale) 6-point-Likert scale: 0 (None) - 1 (Very mild) - 2 (Mild) - 3 (Moderate) - 4 (Strong) - 5 (Very strong). Lower score means a worse outcome.
Evaluate the overall patient's satisfaction. | Day 8
  Assessment by the patient of the overall satisfaction through 5-point Likert scale ((1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied, and 5 = very satisfied)) at Day 8.
Evaluate the overall tolerance of 22‰ Hypertonic seawater solution used as aerosol therapy solution for inhalation. | From Day 1 to Day 7
  Assessment by the investigator of the occurrence of adverse device effect related to the use of 22‰ Hypertonic seawater solution when used as aerosol therapy solution for inhalation.
Evaluate the overall safety of 22‰ Hypertonic seawater solution throughout the study. | From Day 0 to Day 8
  Assessment by the investigators of the occurrence and severity of adverse events (AE)
Evaluate the device related complications rates throughout the study. | From Day 1 to Day 7
  Assessment of the proportion of patients with at least one adverse device effect related to the use of 22‰ Hypertonic seawater solution as an aerosol therapy solution for inhalation .

OTHER OUTCOMES:
Evaluate the performance of 22‰ Hypertonic seawater solution, used as aerosol therapy solution for inhalation, on the evolution of nasal symptom relief using the WURSS-K questionnaire completed by parents for the minor patients of 2 to 3 years old. | At Day 1 and Day 3
  Change in global WURSS-K score as measured in the morning before treatment on Day 1 and Day 3 .
Evaluate the performance of 22‰ Hypertonic seawater solution, used as aerosol therapy solution for inhalation, on the evolution of nasal symptom relief using the WURSS-K questionnaire completed by parents for the minor patients of 2 to 3 years old | Day 1, Day 2, Day 4, Day 5, Day 6, Day 7 and Day 8
  Change in global WURSS-K score as measured in the morning before treatment at Day 2, at Day 4, at Day5, at Day 6, at Day 7 and at Day 8 compared to Day 1 (before treatment) as baseline.
Evaluate the satisfaction of use of the device. | Day 8
  Assessment by the user (patient or patient's parent for minors) of the overall satisfaction of use with a satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Kędzierski, Dr., Principal Investigator — Centrum Medyczne PZU Zdrowie; Michal Tyrek, Dr., Principal Investigator — Centrum Medyczne Pratia Częstochowa
Locations (6):
- Poland (6):
  - Centrum Medyczne Pratia Częstochowa, Częstochowa
  - Centrum Medyczne PZU Zdrowie, Kielce
  - Centrum Medyczne Zdrowie, Kielce
  - Centrum Nowoczesnych Terapii "Dobry Lekarz", Krakow
  - Centrum Medyczne Pratia Poznań, Poznan
  - Krajmed Centrum Medyczne, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided